CLINICAL TRIAL: NCT03982927
Title: Effect of Laparoscopic Skills Workshop on Enhancing Knowledge and Skills of Surgical Residents and Its Comparison With DOPS (Direct Observation of Procedural Skills) Scores - Prospective Cohort Study
Brief Title: Effect of Short Laparoscopic Skills Workshop on Residents' Knowledge and Skills
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Muhammad Rizwan Khan, Associate Professor of Surgery, Aga Khan University
Other Study IDs: 3011-Sur-ERC-14
Record Dates: First submitted 2019-05-26; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Clinical Skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Laparoscopic skills workshop — One day laparoscopic skills workshop was offered to the surgical residents

SUMMARY:
There is no objective data on the outcome of a daylong workshop as commonly offered to the surgical residents by various institutions. Hence we planned a study with the objectives to determine if a one-day laparoscopic skills workshop enhanced the knowledge and skills of surgical residents in minimal access surgery and did the workshop scores have any correlation with the Direct Observation of Procedural Skills (DOPS) scores for the procedures performed in the real life.

The results of our study shall indicate the impact of one-day laparoscopic skills workshop on the knowledge and psychomotor skills of the surgical residents. The skills gained from the workshop shall also be correlated with DOPS scores reflecting the transfer of skills to real life performance.

DETAILED DESCRIPTION:
I. Introduction and Background:

Teaching and learning of psychomotor skills is of paramount importance for surgical residency programs. The 'traditional' model of teaching surgical skills on 'real' patients using graded responsibility is being seriously questioned. More and more focus has recently shifted on the use of models and simulators, with an objective of better preparation of residents for the operating room experience. At Aga Khan University, the focus of surgical training is still on the traditional model, but some innovations have been introduced to enhance the training outcomes and safety of the patients. The innovations include use of short workshops on bench models to train the residents in basic surgical skills before they can operate on the real patients.

The educational impact of such short workshops has been difficult to document, since a long-term follow up is usually not possible. But some recent data suggests that minimal access skills workshops can improve both the knowledge base and motor skills of the trainees. There is also some data to suggest that the skills obtained during a workshop not only have a long lasting effect on the performance of the residents, but may also result in change in practice of the participants. There is no study available where the educational effect of surgical workshop has been correlated with the real time work place based performance of the surgical residents including DOPS (direct observation of procedural skills). DOPS is a form of work place based assessment of residents' knowledge and skills, and can be used as a surrogate marker for the actual performance of the residents in the real world. Improvement of DOPS scores after the workshop might demonstrate the educational influence of the workshop on the residents' knowledge and skills.

II. Rationale and Objective of the Study:

The section of General Surgery at Aga Khan University offers surgical skills workshops to trainees every year to enhance their knowledge and psychomotor skills for the last many years. There is a general perception amongst the trainees and the faculty that these workshops have been quite valuable in refining the skills of the surgical trainees. However, there is no objective data to support this perception and hence there is a need to document the outcome of this important academic activity.

The basic questions that need to be answered are; if there is an effect of laparoscopic skills workshop on enhancing the knowledge and skills of surgical residents and how do the workshop scores correlate with the DOPS (Direct Observation of Procedural Skills) scores. The results of this study may be used for improving the teaching methods for surgical residents as well as the enthusiasm of the faculty involved in such labor intensive activities.

The objective of our study is to determine the difference in the mean scores of knowledge and skills assessment of surgical residents attending the minimal access skills workshop before and after the workshop; and at an interval of 2 months. The second objective is to compare the workshop scores with the DOPS (Direct Observation of Procedural Skills) scores conducted before and after the workshop during the same study period.

III. Methods:

Study Design: This will be a quasi-experimental, single arm, repeat measure study design. The pre-workshop knowledge and skills scores of residents will be compared with immediate post-workshop scores and scores of repeat assessment at 2 months after the workshop. The scores of DOPS on laparoscopic surgery before and after the workshop will also be compared for any change.

Participants: The trainees enrolled in the residency programs of General Surgery and Obstetrics / Gynecology of Aga Khan University have the mandate of acquiring skills of minimal access surgery as a part of their surgical armamentarium. These residents will be invited to participate in the proposed study and the workshop.

Sample Size & Groups: A non-probability, all-inclusive sampling technique will be used. A voluntary participation will be required and the expected number of participants has been estimated to be 30+. The residents will be divided into two groups based on their expected exposure to minimal access surgery Group I: year 1 & 2 residents Group II: year 3, 4 & 5 residents

Setting: The workshop will be a one-day event and conducted at the Anatomy Dissection Hall of the Aga Khan University.

Pre-workshop Assessment:

There will be an MCQs based pre-test to assess the basic knowledge of the residents. The questions will be related to the knowledge of abdominal anatomy, electro-cautery, harmonic scalpel, laparoscopic instruments, port insertion techniques, physiological effects of laparoscopy, complications and management of laparoscopic surgery.

This will be followed by assessment of baseline psychomotor skills of the residents on laboratory-based models. The skills assessed will focus on port insertion, hand-eye coordination and depth perception.

Intervention: The training workshop will consist of didactic lectures, videos and live demonstrations on the basic knowledge and skills related to the minimal access surgery. The components of workshop will include:

1. A lecture focused on introduction to laparoscopic surgery including equipment / instruments, energy sources, operating room setup and team work.
2. Video demonstration of various techniques of creating pneumoperitoneum followed by hands-on practice on bench model.
3. A tutorial on physiological effects, complications and outcome of laparoscopic surgery.
4. Live demonstration of following techniques of minimal access surgery with focus on hand-eye coordination and depth perception, followed by hands-on practice.

   1. Transfer of bean balls across dishes
   2. Passing thread through hooks
   3. Passing rope in graspers / running rope
   4. Cutting a circle on gauze with endo-scissors The various components of the workshop will be spaced by intervals of refreshment and adequate time for hands-on practice to avoid fatigue. (Please see the attached workshop program for time specifications)

Post-workshop Assessment: The workshop will be followed by an immediate post-course assessment consisting of an MCQ test as well as assessment of psychomotor skills on a previously designed preforma.

Interval Assessment: All the participants of the workshop will be asked to keep a log of their involvement in minimal access procedures during the next two months. The purpose of log keeping is to assess their involvement in such procedures which may have an independent effect on their skills as compared to the influence of the workshop alone. At the end of this period, these residents will be invited to an interval assessment of their surgical skills on a previously designed performa to document the durability of surgical skills.

Assessment of Performance: The technical skills of the residents will be video-recorded at all three stages of assessment. The skills will be scored by two independent surgeons using the GOALS scoring system.18 The scores will be compared for inter-rater reliability and any difference will be sorted out by mutual discussion. Surgery residents routinely perform the DOPS and scores will be taken for DOPS performed on minimal access surgery before and after the workshop.

Statistical Analysis: Demographic data will be described in frequencies / percentage, while the pre and post MCQ / skills mean scores (3 readings) will compared by using repeat measures of ANOVA. Pre and post DOPS scores (2 readings) will be compared by using paired t test. The scores of MCQs, skills and DOPS will be compared by using correlation coefficient (Pearson r).

The effect of year of residency on scores will be analyzed by using one way ANOVA. Construct validity of the intervention will be calculated by comparing the scores of various years / level of experience. Inter-rater reliability of assessors will be assessed by comparing the scores of two assessors (Bald Altman test).

Ethical Clearance: An ethical approval for the conduct of the study will be obtained from the institutional ethics committee. An informed consent will be obtained from the participants for inclusion in the study.

IV. Results:

The detailed results will be given after completion of the study. It is expected that post-workshop knowledge and assessment scores of surgical residents will be better as compared to pre-workshop scores. The performance of residents in DOPS will also improve after the workshop. It is also expected that the scores of the senior residents will be better than the junior residents.

V. Conclusions:

The results of the study will objectively establish the effect of surgical skills workshop on enhancing the knowledge and skills of the surgical residents. Te study will also demonstrate the correlation between the workshop and DOPS scores.

ELIGIBILITY:
Inclusion Criteria:

* All general surgery and gynaecology residents were invited for participation in the study

Exclusion Criteria:

* Any resident who refused voluntary participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A non-probability, all-inclusive sampling technique was used. The total number of participants recruited for this study was 33, including 24 residents from General Surgery and 9 residents from Obstetrics & Gynaecology. For subgroup analysis, the residents were divided into two groups based on their expected exposure to minimal access surgery:
  Group I: year 1 & 2 residents Group II: year 3, 4 & 5 residents
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Cognitive Skills | 02 months
  MCQ sores before and after the workshop; minimum score: zero; maximum score: 30
Clinical Skills | 03 months
  GOALS (global operative assessment of laparoscopic skills) scale for assessment of clinical skills in laparoscopy. This is a validated tool and has 5 parameters assessed on a Likert scale of 1 to 5. Higher the score, better the value.

SECONDARY OUTCOMES:
Clinical Skills (in real life) | 06 months
  Comparison of Direct Observation of Procedural skills (DOPS) Scores before and after the workshop. This is a validated tool used for assessment of procedural skills. It has a number of parameters assessed on a Likert scale of 1 to 3. Higher the score, better the value.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data

REFERENCES:
- [Derived] Khan MR, Shariff AH, Nasim S, Sayyed RH, Effendi MS, Pinjani S. Effectiveness of Laparoscopic Skills Workshop on Enhancing Knowledge and Skills of Surgical Residents and Its Comparison with DOPS (Direct Observation of Procedural Skills) Scores: Prospective Cohort Study. Med Sci Educ. 2020 May 6;30(2):861-867. doi: 10.1007/s40670-020-00966-5. eCollection 2020 Jun. PMID 34457743